CLINICAL TRIAL: NCT03900026
Title: A Randomized Trial of Evolocumab on Saphenous Vein Graft Patency Following Coronary Artery Bypass Surgery (NEWTON-CABG)
Brief Title: Effect of Evolocumab on Saphenous Vein Graft Patency Following Coronary Artery Bypass Surgery
Acronym: NEWTON-CABG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Applied Health Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NEWTON CABG (CardioLink-5)
Record Dates: First submitted 2019-03-28; First posted 2019-04-02 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-05

CONDITIONS: Coronary Artery Bypass Graft Surgery; Atherosclerosis; Vein Occlusion
Keywords: Coronary Artery Bypass Surgery; CABG; Saphenous Vein Graft; Evolocumab; Repatha
MeSH Terms: conditions — Atherosclerosis | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: Multicenter, double-blind, randomized, placebo-controlled, parallel group study of evolocumab.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo Treatment (Placebo Comparator): Participants will receive subcutaneous injections of the placebo Q2W (every 2 weeks)
  Interventions: Other: Placebo
- Evolocumab Treatment (Experimental): Participants will receive subcutaneous injections of 140mg of evolocumab Q2W (every two weeks)
  Interventions: Drug: Evolocumab

INTERVENTIONS:
Drug: Evolocumab — REPATHA (evolocumab) is a human immunoglobulin G2 (IgG2) monoclonal antibody that has high affinity binding to Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9); it will be administered via subcutaneous injection
  Other Names: Repatha®
  Arms: Evolocumab Treatment
Other: Placebo — Placebo cartridges will contain vehicle only; placebo will be administered via subcutaneous injection.
  Other Names: Control
  Arms: Placebo Treatment

SUMMARY:
The purpose of this study is to determine if evolocumab added to regular statin therapy improves vein graft patency after coronary artery bypass graft (CABG) surgery.

DETAILED DESCRIPTION:
Coronary artery bypass graft (CABG) surgery is a procedure in which an artery or vein from the body is grafted to a critically narrowed coronary artery to restore flow of oxygenated blood to the heart. Statins are frequently prescribed after CABG surgery in order to lower LDL cholesterol levels and reduce the chances of coronary artery obstruction recurring. Despite this preventive measure, new vein grafts do end up becoming blocked in a significant proportion of patients. Evolocumab (Repatha®) is a recently approved medication that has been shown to effectively lower LDL cholesterol levels in the blood.

NEWTON-CABG is an investigator-initiated multicenter, double-blind, randomized, placebo-controlled, parallel group study of evolocumab [140mg administered subcutaneously (SC) every two weeks (Q2W)] added to statin therapy for 24 months postoperatively in a broad population of patients undergoing CABG surgery. Eligible subjects will be randomized to receive evolocumab or placebo within 21 days of index CABG. Prior to randomization, post-operative patients will be on moderate or high intensity statin therapy (atorvastatin 40-80mg, rosuvastatin 20-40mg or simvastatin 40mg daily unless another statin/dose or non-statin alternative is clinically justified). A CTAngiogram will be conducted at 24 months following CABG. Routine study visits will be done 3, 6, 12, 18 and 24 months post-surgery.

This study is supported by Amgen Inc.

ELIGIBILITY:
Inclusion Criteria - To be considered eligible for participation in this study, a participant must satisfy each of the following criteria:

1. Age ≥ 18 years
2. Scheduled to undergo coronary artery bypass graft (CABG) surgery (with or without cardiopulmonary bypass (CPB); with or without single valve repair/replacement)
3. CABG procedure included/planned to include at least two saphenous vein grafts
4. CABG procedure occurred within the past 21 days, or is planned within the next 60 days
5. On a moderate to high intensity statin therapy (defined as atorvastatin 40-80mg daily, rosuvastatin 20-40mg or simvastatin 40mg daily) unless a lower dose, or another statin or non-statin therapy is clinically justified

Exclusion Criteria - A participant will be ineligible for participation in this study if he or she satisfies any one or more of the following criteria:

1. Patients in whom additional lowering of LDL-C with evolocumab is deemed to be clinically inappropriate
2. Allergy to contrast dye
3. Known severe hepatic impairment (Childs-Pugh, Class C).
4. Known renal disease with estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73m2
5. Recipient of any major organ transplant (eg, lung, liver, heart, bone marrow)
6. Use of cholesterylester transfer protein (CETP) inhibition treatment within 12 months prior to randomization.
7. Current, prior within past year, or known planned use of PCSK9 inhibition treatment
8. Severe cardiovascular or concomitant non-cardiovascular disease that is expected to reduce life expectancy to less than 2 years
9. Major active infection, or major hematologic, renal, respiratory, metabolic, gastrointestinal or endocrine dysfunction
10. Women who are pregnant or breastfeeding
11. Women of child bearing potential who are unwilling to use proper family planning or birth control methods to avoid pregnancy. Women are considered post-menopausal and not of childbearing potential after 12 months of natural (spontaneous) amenorrhea or have had a surgical procedure such as hysterectomy which makes pregnancy impossible.
12. Known intolerance or allergy to evolocumab or other PCSK9 inhibitors.
13. Currently taking simvastatin >40mg/day, niacin or bile acid sequestrants
14. Known latex allergy
15. Inability to comply with protocol-required study visits or procedures, including administration of study drug
16. Known history of cancer within the past 5 years (except for carcinoma in-situ of the cervix, stage 1 prostate cancer or adequately treated non-melanoma carcinomas of the skin)
17. Participation in another investigational device or drug study which is likely to affect the primary outcome, within 30 days of planned initiation of study drug
18. NYHA class IV
19. Pacemaker or other implantable device implanted within 30 days prior to screening

Additional postoperative exclusion criteria:

1. Received only <2 vein grafts
2. Major peri-operative complications following CABG surgery (e.g. stroke, MI, renal failure requiring dialysis, or postoperative ICU stay > 5 days) prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 782 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Saphenous vein graft disease rate (VGDR) | 24 months post CABG
  Saphenous vein graft disease rate (VGDR) is defined as the proportion of vein grafts with significant stenosis or total occlusion (≥50%) on 64-slice (or greater) cardiac CT angiography (CTA) or clinically indicated coronary angiography.

SECONDARY OUTCOMES:
The proportion of patients with at least 1 vein graft totally (100%) occluded. | 24 months post CABG
  Proportion of patients who have at least 1 totally (100%) occluded vein graft at 24 months post CABG.
The percentage of vein grafts which are totally (100%) occluded grafts. | 24 months post CABG
  Percentage of vein grafts that are totally (100%) occluded at 24 months post CABG.
Hierarchical composite of the following (each assessed by total wins for each treatment group and the win ratio): | 24 months post CABG
  1. time to cardiovascular death from baseline to end of study
  2. time to first myocardial infarction from baseline to end of study
  3. time to first coronary revascularization from baseline to end of study
  4. number of vein grafts with 100% stenosis at end of study
  5. number of vein grafts with 50-99% stenosis at end of study
  6. number of occluded arterial grafts at end of study
  7. total plaque volume at end of study
  a. time to cardiovascular death from baseline to end of study b. time to first myocardial infarction from baseline to end of study c. time to first coronary revascularization from baseline to end of study d. number of vein grafts with 100% stenosis at end of study e. number of vein grafts with 50-99% stenosis at end of study f. number of occluded arterial grafts at end of study g. total plaque volume at end of study

OTHER OUTCOMES:
Composite rate of fatal and non-fatal myocardial infarction, fatal and non-fatal stroke, cardiovascular death, coronary heart disease death, repeat coronary revascularization | 24 months post CABG
  composite rate of occurrence of the above mentioned clinical outcomes at 24 months post CABG.
Rate of fatal and non-fatal myocardial infarction. | 24 months post CABG
  Rate of occurrence of the above mentioned clinical outcome at 24 months post CABG.
Rate of fatal and non-fatal stroke. | 24 months post CABG
  Rate of occurrence of the above mentioned clinical outcome at 24 months post CABG.
Rate of cardiovascular death. | 24 months post CABG
  Rate of occurrence of the above mentioned clinical outcome at 24 months post CABG.
Rate of coronary heart disease death. | 24 months post CABG
  Rate of occurrence of the above mentioned clinical outcome at 24 months post CABG.
Rate of repeat coronary revascularization. | 24 months post CABG
  Rate of occurrence of the above mentioned clinical outcome at 24 months post CABG.
Rate of all-cause mortality. | 24 months post CABG
  Proportion of patients who have died at 24 months post CABG.
Rate of total vein graft patency at 24 months. | 24 months post CABG
  Rate of total vein graft patency defined as 1-VGDR at 24 months post CABG.
Percentage of patients free of vein graft disease at 24 months. | 24 months post CABG
  Percentage of patients who are free of vein graft disease at 24 months defined as having no vein grafts with ≥ 50% stenosis.
Vein graft plaque volume. | 24 months post CABG
  Volume of vein graft plaque at 24 months post CABG.

CONTACTS AND LOCATIONS:
Overall Officials: David Mazer, MD, Principal Investigator — Unity Health Toronto; Subodh Verma, MD, Principal Investigator — Unity Health Toronto; Lawrence Leiter, MD, Study Chair — Unity Health Toronto
Locations (22):
- United States (5):
  - San Francisco VA Medical Center, San Francisco, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Maine Medical Center, Portland, Maine
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
- Australia (4):
  - Royal Adelaide Hospital, Adelaide
  - Flinders Medical Centre, Bedford Park
  - Monash University, Melbourne
  - Fiona Stanley Hospital, Murdoch
- Canada (10):
  - University of Alberta, Edmonton, Alberta
  - New Brunswick Heart Centre, Saint John's, New Brunswick
  - Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - One Heart Care, Mississauga, Ontario
  - North York Diagnostic and Cardiology Centre, North York, Ontario
  - Sunnybrook Health Sciences Center, North York, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec
  - Foothills Medical Centre, Calgary
- Hungary (3):
  - Medical Centre Hungarian Defence Forces, Budapest
  - Semmelweis University Heart and Vascular Centre, Budapest
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Verma S, Leiter LA, Teoh H, Mancini GBJ, Quan A, Elituv R, Verma M, Misner E, Szarek M, Thorpe KE, Saha T, Whitlock RP, Yanagawa B, Merkely B, Juni P, Koren MJ, Nicholls SJ, Bhatt DL, Mazer CD. Effect of evolocumab on saphenous vein graft patency after coronary artery bypass surgery (NEWTON-CABG CardioLink-5): an international, randomised, double-blind, placebo-controlled trial. Lancet. 2025 Sep 20;406(10509):1223-1234. doi: 10.1016/S0140-6736(25)01633-2. Epub 2025 Sep 1. PMID 40907505